CLINICAL TRIAL: NCT03841604
Title: A Randomised, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Safinamide 100mg Once Daily, as add-on Therapy, in Idiopathic Parkinson's Disease (PD) Patients With Motor Fluctuations and PD Related Chronic Pain
Brief Title: Effect of Safinamide on Parkinson's Disease Related Chronic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z7219M01; 2017-002426-20 (EudraCT Number)
Record Dates: First submitted 2019-01-30; First posted 2019-02-15 (Actual); Results first posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2020-05

CONDITIONS: Idiopathic Parkinson Disease
Keywords: Parkinson disease; Safinamide
MeSH Terms: conditions — Parkinson Disease | interventions — safinamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Safinamide methanesulfonate film coated tablets once daily, 50 mg and 100 mg. Safinamide methanesulfonate 50 mg and 100 mg tablets was administered orally, OD, with or without food, at breakfast time when the subject was taking their morning dose of L-DOPA.
  Subjects received study drug 50 mg (from Day 1 to Day 7) and then 100 mg (from Day 8 onwards). The dose of 100 mg/day (titrated from 50 mg/day after 1 week) was selected based on the results of previous studies in patients with PD and from the results of a post hoc analysis that investigated the effects of safinamide on pain.
  Interventions: Drug: Safinamide Methanesulfonate
- Placebo (Placebo Comparator): Safinamide methanesulfonate matching placebo film coated tablets once daily. The matching placebo was administered orally, OD, in tablets, with or without food, at breakfast time when the subject was taking their morning dose of L-DOPA.
  Interventions: Other: Safinamide methanesulfonate matching placebo

INTERVENTIONS:
Drug: Safinamide Methanesulfonate — 50 mg, 100 mg
  Other Names: Xadago
  Arms: Experimental
Other: Safinamide methanesulfonate matching placebo — 50 mg, 100 mg
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Primary objective:

• To evaluate the potential efficacy of safinamide 100 mg once daily (OD), compared with placebo, as add-on therapy for PD-related chronic pain

Secondary objectives:

* Percentage of pain responders
* Clinical Global Impression for pain
* Patient Global Impression for pain
* Reduction in use of pain drugs
* Mood
* Motor and non-motor symptoms

Safety Objectives:

• Safety and tolerability

DETAILED DESCRIPTION:
This is a Phase IV, international, multicentre, randomised, double-blind, placebo controlled study in idiopathic Parkinson's disease (IPD) patients, experiencing motor fluctuations and PD-related chronic pain while on stable doses of levodopa (L-Dopa), to Evaluate the Efficacy and Safety of Safinamide 100 mg Once Daily, as Add-On Therapy.

The study consisted of:

* A screening period of up to 1 to 2 weeks.
* A treatment period of 16 weeks.
* A telephone follow-up call at 1 week after the end of treatment. Eligible subjects were randomly assigned in a ratio of 2:1 to receive either safinamide (50 mg or 100 mg) or matching placebo. At Day 1, eligible subjects entered the treatment period to receive safinamide 50 mg (from Day 1 to Day 7) and then 100 mg (from Day 8 onwards) orally OD. After completion of all baseline assessments, subjects received the first dose of study drug at the study center and, thereafter, study drug was to be taken at home each morning along with their first morning dose of L-DOPA and other (if any) PD medications. On Day 8, the dose of study drug was increased, at home, to 100 mg OD. Each subject received treatment for 16 weeks, with visits at Week 0/Day 1 (baseline) and at Weeks 4, 8, and 16 (or early termination). From Day 1 onwards, subjects recorded the use of as-needed (PRN) medications along with indicating the worst pain they experienced on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 30 years of age or older, at the time of signing the informed consent.
2. Diagnosed with IPD by using the United Kingdom Parkinson's Disease Society Brain Bank criteria for more than 5 years duration.
3. Receiving treatment with a stable dose of oral L-Dopa (including controlled release [CR], immediate release [IR] or a combination of CR/IR), with and without benserazide/carbidopa, with or without addition of a catechol O-methyltransferase (COMT) inhibitor and may be receiving concomitant treatment with stable doses of a dopamine agonist, an anticholinergic and/or amantadine for at least 4 weeks prior to the randomisation (baseline visit).
4. Hoehn and Yahr stage between 2-3 (inclusive) during the "ON" phase at the screening visit.
5. Experiencing motor fluctuations following optimum titration of treatment medications and within the 4 weeks immediately prior to randomisation.
6. Experiencing chronic pain (i.e. ongoing for ≥3 months prior to screening visit); the Investigator must consider chronic pain directly related to PD and not explained by any other health problem (e.g. peripheral neuropathy, organ disease or arthritis pain) OR consider the intensity of chronic pain specifically aggravated by PD.
7. If taking regular analgesics, the treatment regimen should be stable in the 4 weeks prior to the randomisation visit.
8. Able to maintain an accurate and complete electronic diary with the help of a caregiver.
9. Male or female

   •A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: i.Not a woman of childbearing potential (WOCBP) OR ii.A WOCBP who agrees to follow the contraceptive guidance
10. Capable of giving signed informed consent

Exclusion Criteria:

1. Any form of Parkinsonism other than IPD.
2. Diagnosis of chronic migraine (>15 days per month) or cancer pain.
3. History of bipolar disorder, depression, schizophrenia or other psychotic disorder requiring treatment with neuroleptics.
4. History of dementia or cognitive dysfunction.
5. Severe, peak dose or biphasic dyskinesia.
6. Unpredictable or widely swinging fluctuations.
7. Ophthalmologic history including any of the following conditions: albinism, uveitis, retinitis pigmentosa, retinal degeneration, active retinopathy, severe progressive diabetic retinopathy, inherited retinopathy or family history of hereditary retinal disease.
8. Moderate or severe liver failure using the Child-Pugh classification score.
9. History of drug and/or alcohol abuse within 12 months prior to screening as defined by the current edition of the Diagnostic and Statistical Manual of Mental Disorders.
10. Allergy/sensitivity, intolerance or contraindications to Safinamide.
11. Treatment with monoamine oxidase inhibitors (MAOIs), levodopa infusion, pethidine, fluoxetine, fluvoxamine less than 4 weeks prior to the randomisation visit
12. Use of any investigational drug or device within 30 days prior to screening or 5 half-lives, whichever is the longest
13. Previous treatment with Safinamide in the 9 months before the screening visit
14. Mini-Mental State Exam (MMSE) total score <24 at screening.
15. NRS score ≤ 4 points at randomization visit.
16. Any clinically significant condition which, in the opinion of the Investigator, would not be compatible with study participation or represent a risk for participants while in the study

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Keywood, MD, Study Director — Zambon SpA
Locations (45):
- Austria (2):
  - Medizinische Universitat Innsbruck, Innsbruck
  - Institut für Neuroimmunologische und Neurodegenerative Erkrankungen, Vienna
- France (6):
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - CHU de GRENOBLE, Grenoble
  - Hopitaux de La Timone, Marseille
  - Centre Hospitalier Universitaire de Nimes, Nîmes
  - Hopital de Hautepierre, Strasbourg
  - Hôpital Pierre-Paul Riquet, Toulouse
- Germany (10):
  - St. Joseph Krankenhaus Berlin, Berlin
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Katholische Kliniken Ruhrhalbinsel GmbH, Essen
  - Neurologische Praxis, Gera
  - University Medicine Göttingen Germany, Göttingen
  - Klinik Haag i. OB, Haag
  - Universitätsklinikum Gießen und Marburg GmbH, Marburg
  - Universitätsklinikum Münster, Münster
  - NeuroPoint Akademie, Ulm
  - Universitätsklinikum Ulm, Ulm
- Italy (11):
  - Zambon Investigative Site, Chieti
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Centro per la Malattia di Parkinson e i Disturbi del Movimento, Milan
  - Ospedale San Raffaele S.r.l. - PPDS, Milan
  - Azienda Ospedaliera Di Perugia, Perugia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Istituto Neurologico Mediterraneo Neuromed, Pozzilli
  - Fondazione PTV Policlinico Tor Vergata, Roma
  - Ospedale San Giovanni Battista - ACISMOM, Roma
  - IRCCS San Raffaele Pisana, Roma
  - Azienda Ospedaliera Universitaria OO.RR. San Giovanni di Dio Ruggi d'Aragona, Salerno
- Spain (16):
  - Hospital del Mar, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebrón - PPDS, Barcelona
  - C.A.U de Burgos - Hospital Universitario de Burgos, Burgos
  - Hospital Puerta del Mar, Cadiz
  - Hospital Universitario de Donostia, Donostia / San Sebastian
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Madrid
  - Hospital HM Puerta del Sur, Móstoles
  - Clinica Universidad Navarra, Pamplona
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 94 subjects were enrolled in the study; 46 subjects were randomly assigned to safinamide and 25 subjects to placebo. Overall, 23 subjects were screen failures.
  Overall, 60 subjects (83.3%) completed the study, and 11 subjects discontinued from the study.
Period: Overall Study
Arm/Group | Experimental | Placebo
Started | 46 | 25
Completed | 38 | 22
Not Completed | 8 | 3
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Adverse Event | 4 | 2
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set: all randomised subjects assigned to study intervention and who took at least 1 dose of study intervention.
Groups:
- Experimental: Safinamide methanesulfonate film coated tablets once daily
  Safinamide Methanesulfonate: 50 mg, 100 mg
- Placebo: Safinamide methanesulfonate matching placebo film coated tablets once daily
  Safinamide methanesulfonate matching placebo: 50 mg, 100 mg
- Total: Total of all reporting groups
Arm/Group | Experimental | Placebo | Total
Number analyzed (Participants) | 46 | 25 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 11 | 30
  >=65 years | 27 | 14 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (10.55) | 66.4 (11.82) | 66.3 (10.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 12 | 37
  Male | 21 | 13 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 44 | 24 | 68
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 16 in Pain Severity (NRS-11 Scale) - Full Analysis Set
Description: To evaluate the potential efficacy of safinamide 100 (mg od), compared to placebo, as add-on therapy, for change pain severity ("average worst pain experienced in the last 7 days"), as assessed by an 11-point Numerical Rating Scale (NRS). Based on this scale, 0 point is the minimum and 10 point is the maximum. The higher the score, the more severe the pain.
Time Frame: Baseline and Week 16
Population: Full Analysis Set:All randomized subjects in the study, with at least one measurement of the primary efficacy variable following at least one dose of study drug. Please note that n (39 and 20) above reported is the number of subjects with observed average worst pain score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 39 | 20
score on a scale | -1.6 (2.01) | -0.8 (1.29)
Statistical Analysis 1: Comparison: Experimental vs Placebo; Test type: Superiority; p = 0.1695, Mixed Model Repeated Measures; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.75 to 0.32], Standard Error of Mean 0.52

2. Primary Outcome: Change From Baseline to Week 16 in Pain Severity (NRS-11 Scale) - Per Protocol Set
Description: as for outcome 1
Time Frame: Baseline and Week 16
Population: Per Protocol Set : The PP set was a subset of subjects in the FAS who completed the study and for whom no relevant protocol deviations were documented
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 35 | 19
score on a scale | -1.6 (2.05) | -0.8 (1.33)
Statistical Analysis 1: Comparison: Experimental vs Placebo; Test type: Other; p = 0.0784, Mixed Model Repeated Measures; Least square mean difference = -1, 95% CI 2-sided [-2.1 to 0.12], Standard Error of Mean 0.55

3. Secondary Outcome: Number of Subjects With a Reduction of ≥2 Points in Pain Severity at Week 16, Compared to Baseline
Description: Reduction in pain severity (based on the "average worst pain experienced in the last 7 days") of ≥ 2 points was assessed by an 11-point NRS (numerical rating scale), compared to baseline. Based on this scale, 0 point is the minimum and 10 point is the maximum. The higher the score, the more severe the pain.
Time Frame: Week 16
Population: Full Analysis Set: All randomized subjects in the study, with at least one measurement of the primary efficacy variable following at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 45 | 23
Participants | 15 | 3
Statistical Analysis 1: Comparison: Experimental vs Placebo; Test type: Other; p = 0.0744, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.23, 95% CI 2-sided [-0.45 to -0.01]

4. Secondary Outcome: The Change From Baseline to Week 16 in the Clinical Global Impression of Change (CGI-C) Score for Pain
Description: CGI-C (Clinical Global Impression - Change) score for pain is a seven-point scale that indicates the patient's impression of change for relevant symptoms. It ranges from "substantial improvement" to "substantial worsening":
  1. = substantial improvement;
  2. = moderate improvement;
  3. = minimum improvement;
  4. = No change;
  5. = Minimum worsening;
  6. = moderate worsening;
  7. = substantial worsening. of course the higher the score, the worse the outcome.
Time Frame: Baseline and Week 16
Population: Full Analysis Set: Full Analysis Set: All randomized subjects in the study, with at least one measurement of the primary efficacy variable following at least one dose of study drug. Please note that n above reported (37 and 20) is the number of subjects with observed CGI-C score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 37 | 20
score on a scale | 3.4 (1.09) | 3.5 (1.00)
Statistical Analysis 1: Comparison: Experimental vs Placebo; Test type: Other; p = 0.7247, Mixed Model Repeated Measures; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.70 to 0.49], Standard Error of Mean 0.30

5. Secondary Outcome: The Global Impression of Severity (CGI-S) Score for Pain at Week 16
Description: The CGI-S (Clinical Global Impression - Severity) score is a seven-point scale which asks the clinician one question: "considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated as follow:
  1. = normal, not at all ill;
  2. = borderline mentally ill;
  3. = mildly ill;
  4. = moderately ill;
  5. = markedly ill;
  6. = severely ill;
  7. = among the most severely ill patients. of course the higher the score, the worse the outcome.
Time Frame: Baseline and Week 16
Population: Full Analysis Set: All randomized subjects in the study, with at least one measurement of the primary efficacy variable following at least one dose of study drug. Please note that n (44 and 22) here reported is the number of subjects with observed CGI-S score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 44 | 22
score on a scale
  Baseline | 3.8 (0.65) | 3.8 (0.66)
  Week 16: number analyzed (Participants) | 37 | 20
  Week 16 | 3.4 (0.76) | 3.5 (0.76)
Statistical Analysis 1: Comparison: Experimental vs Placebo; Test type: Other; p = 0.9052, Mixed Model Repeated Measures; Mean Difference (Net) = -0.0, 95% CI 2-sided [-0.43 to 0.38], Standard Error of Mean 0.20

6. Secondary Outcome: The Change From Baseline to Week 16 in the Patient Global Impression of Change (PGI-C) Score for Pain
Description: The Patients' Global Impression of Change (PGI-C) scale is designed to capture the subject's perception of change in activity limitations, symptoms, emotions, an overall quality of life. These areas are captured using a 7- point scale, indicating:
  1. = no change (or condition has got worse);
  2. = almost the same, hardly any change at all;
  3. = a little better, but not noticeable change;
  4. = somewhat better, but the change has not made any real difference;
  5. = moderately better, and a slight but noticeable change;
  6. = better and a definite improvement that has made a real and worthwhile difference;
  7. = a great deal better, and a considerable improvement that has made all the difference.
  Of course, the higher the score, the better the outcome.
Time Frame: Baseline and Week 16
Population: Full Analysis Set: All randomized subjects in the study, with at least one measurement of the primary efficacy variable following at least one dose of study drug. Please note that n (33 and 20) here reported is the number of subjects with observed PGI-C score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 33 | 20
score on a scale | 2.7 (1.33) | 2.5 (1.28)
Statistical Analysis 1: Comparison: Experimental vs Placebo; Test type: Other; p = 0.7115, Mixed Model Repeated Measures; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.61 to 0.88], Standard Error of Mean 0.37

7. Secondary Outcome: Number of Subjects With Concomitant Use of Pain Drugs at Different Timepoints
Description: This outcome describes the number of subjects which had concomitant assumption of pain drugs at different timepoints.
Time Frame: Baseline, weeks 4, 8 and 16
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 45 | 23
participants
  Subjects with Concomitant Pain Drug at baseline | 0 | 0
  Subjects with Concomitant Pain Drug at week 4 | 0 | 1
  Subjects with Concomitant Pain Drug at week 8 | 0 | 0
  Subjects with Concomitant Pain Drug at week 16 | 0 | 0
Statistical Analysis 1: Comparison: Experimental vs Placebo; Test type: Superiority; p = 0.1967, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.04, 95% CI 2-sided [-0.04 to 0.12]

8. Secondary Outcome: Amount of PRN PD Pain Medication: Count of Subjects Who Used PRN PD Pain Medication in the 7 Days Preceding Visits
Description: Total count of patients who used PRN (meaning "when necessary") Parkinson's Disease Pain Medications was expressed both in number and in percentage.
  The analysis of amount of concomitant PRN PD pain medications as reported in the subject diary was summarized:
  * as the number of subjects who were taking pain medication in the 7 days preceding visits at different timepoints;
  * in the number of days on which PRN PD pain medication was taken at different timepoints.
Time Frame: at Baseline and weeks 4, 8 and 16
Population: Full Analysis Set:All randomized subjects in the study, with at least one measurement of the primary efficacy variable following at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 45 | 23
Participants
  Subjects with PRN PD Pain Medication at Baseline | 12 | 7
  Subjects with PRN PD Pain Medication at week 4 | 8 | 5
  Subjects with PRN PD Pain Medication at week 8 | 5 | 4
  Subjects with PRN PD Pain Medication at week 16 | 5 | 4
Statistical Analysis 1: Comparison: Experimental vs Placebo; Test type: Superiority; p = 0.5122, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.06, 95% CI 2-sided [-0.13 to 0.26]

9. Secondary Outcome: Amount of PRN PD Pain Medication: Number of Days on Which PRN PD Pain Medication Was Taken at Different Timepoints
Description: The analysis of amount of concomitant PRN PD pain medications as reported in the subject diary was summarized:
  * as the number of days on which PRN PD pain medication was taken at different timepoints.
  * as the number of subjects who were taking pain medication in the 7 days preceding visits at different timepoints.
Time Frame: At Baseline and weeks 4, 8 and 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: number of days
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 27 | 19
number of days
  Baseline: number analyzed (Participants) | 11 | 7
  Baseline | 3.2 (2.44) | 4.1 (2.34)
  week 4: number analyzed (Participants) | 8 | 4
  week 4 | 4.8 (2.76) | 4.3 (3.20)
  week 8: number analyzed (Participants) | 4 | 4
  week 8 | 6.0 (2.00) | 4.5 (1.00)
  week 16: number analyzed (Participants) | 4 | 4
  week 16 | 4.5 (1.73) | 5.3 (1.71)

10. Secondary Outcome: Change From Baseline to Week 16 in the Hospital Anxiety and Depression Scale (HADS) Score
Description: The Hospital Anxiety and Depression Scale (HADS) was devised to measure anxiety and depression in a general medical population of patients through a unique questionnaire which takes 2-5 min to be completed. The questionnaire consists of a total of 14 items: seven items for the anxiety subscale (HADS Anxiety) and seven items for the depression subscale (HADS Depression). HADS Anxiety focus mainly on symptoms of generalized anxiety disorder and HADS Depression is focused on anhedonia, the main symptom of depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for anxiety subscale and the same for depression subscale, where:
  0-7 = Normal 8-10 = Borderline abnormal (borderline case). 11-21 = Abnormal (case) The two subscores are then summed up to obtain a total Hospital Anxiety and Depression Scale (HADS). The total scale range is 0-42. The higher the score, the worse the anxiety/depression status.
Time Frame: Baseline and Week 16
Population: Full Analysis Set: All randomized subjects in the study, with at least one measurement of the primary efficacy variable following at least one dose of study drug. Please note that n (33 and 20) is the number of subjects with observed HADS score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 33 | 20
score on a scale | -1.5 (6.03) | -2.0 (4.36)
Statistical Analysis 1: Comparison: Experimental vs Placebo; Test type: Other; p = 0.7376, ANCOVA; Mean Difference (Net) = -0.4, 95% CI 2-sided [-3.03 to 2.16], Standard Error of Mean 1.29

11. Secondary Outcome: The Change From Baseline to Week 16 in MDS-UPDRS
Description: Change in the MDS-UPDRS = Movement Disorder Society-Unified Parkinson's Disease Rating Scale The MDS-UPDRS is defined by 4 Parts, each composed by a different number of items. Each item is rated on a 5-point Likert-type scale (ranging from 0 to 4); Part I (non-motor experiences of daily living; 13 items) Part II (motor experiences of daily living;13 items) Part III (motor examination; 33 items) Part IV (motor complications; 6 items) The MDS-UPDRS has a minimum score of 0 and a maximum score of 260. The higher the score, the more severe the impairment.
Time Frame: Baseline and Week 16
Population: Full Analysis Set: All randomized subjects in the study, with at least one measurement of the primary efficacy variable following at least one dose of study drug. Please note that n (31 and 19) is the number of subjects with observed MDS-UPDRS score
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 31 | 19
score on a scale | -6.8 (13.79) | -4.8 (11.68)
Statistical Analysis 1: Comparison: Experimental vs Placebo; Test type: Other; p = 0.5349, Mixed Model Repeated Measures; Mean Difference (Net) = -2.5, 95% CI 2-sided [-10.33 to 5.43], Standard Error of Mean 3.92

ADVERSE EVENTS:
Time Frame: Adverse events were collected Up to 14 days before Day 1 (Screening period), at baseline, at week 4-8-16 and at follow up period, up to 19 weeks.
Description: Please note that TEAEs were reported in the CSR for safinamide (whichever was the dose) and placebo, separately.
  No differenciacion between IMP doses for TEAE was done, nor is available.
Arm/Group | Experimental | Placebo
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/46 | 2/25
Other Adverse Events (participants affected / at risk) | 19/46 | 12/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=46) | Placebo (N=25)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Lacunar Infarction (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=46) | Placebo (N=25)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Pterygium (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dyskinesia (Nervous system disorders) | 2 (2) | 0 (0)
Hyperkinesia (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Motor dysfunction (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT03841604/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/04/NCT03841604/SAP_001.pdf